CLINICAL TRIAL: NCT00636610
Title: A Randomized, Placebo-Controlled Phase II Study of Vismodegib (GDC-0449, Systemic Hedgehog Antagonist) With Concurrent Chemotherapy and Bevacizumab As First-Line Therapy for Metastatic Colorectal Cancer
Brief Title: A Study of Vismodegib (GDC-0449, Hedgehog Pathway Inhibitor) With Concurrent Chemotherapy and Bevacizumab As First-Line Therapy for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHH4429g
Record Dates: First submitted 2008-03-05; First posted 2008-03-14 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Hedgehog; CRC; Colorectal Cancer; Hedgehog Pathway Inhibitor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HhAntag691; Bevacizumab; IFL protocol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vismodegib 150 mg (Experimental): Patients received vismodegib 150 mg orally once daily starting on Day 3 of each 2-week treatment cycle. In addition, patients received either Modified FOLFOX (FOL=leucovorin calcium [folinic acid], F=fluorouracil, OX=oxaliplatin) + bevacizumab or FOLFIRI (FOL=leucovorin calcium [folinic acid] F=fluorouracil, IRI=irinotecan hydrochloride) + bevacizumab on Days 1-3 of each 2-week treatment cycle. The decision of which regimen (FOLFOX or FOLFIRI) to use was made by the treating physician and patient.
  Interventions: Drug: Vismodegib 150 mg; Drug: Bevacizumab; Drug: Modified FOLFOX; Drug: FOLFIRI
- Placebo to vismodegib (Placebo Comparator): Patients received placebo to vismodegib orally once daily starting on Day 3 of each 2-week treatment. In addition, patients received either Modified FOLFOX (FOL=leucovorin calcium [folinic acid], F=fluorouracil, OX=oxaliplatin) + bevacizumab or FOLFIRI (FOL=leucovorin calcium [folinic acid] F=fluorouracil, IRI=irinotecan hydrochloride) + bevacizumab on Days 1-3 of each 2-week treatment cycle. The decision of which regimen (FOLFOX or FOLFIRI) to use was made by the treating physician and patient.
  Interventions: Drug: Placebo to vismodegib; Drug: Bevacizumab; Drug: Modified FOLFOX; Drug: FOLFIRI

INTERVENTIONS:
Drug: Vismodegib 150 mg — Vismodegib 150 mg was provided in hard gelatin capsules in 3 different strengths, 25 mg, 125 mg, and 150 mg.
  Other Names: GDC-0449; Erivedge
  Arms: Vismodegib 150 mg
Drug: Placebo to vismodegib — Placebo to vismodegib consisted of the excipients for vismodegib without the active molecule in hard gelatin capsules matching the active drug product in color and size.
  Arms: Placebo to vismodegib
Drug: Bevacizumab — Bevacizumab 5 mg/kg was administered intravenously (IV) over 90 minutes for the first infusion, shortening to 60 and 30 minutes for subsequent infusions.
Drug: Modified FOLFOX — Following administration of bevacizumab, patients received oxaliplatin 85 mg/m^2 IV administered over 90 minutes concurrently with folinic acid 400 mg/m^2 (d,I-racemic form, or 200 mg/m^2 I-isomer form) IV administered over 120 minutes, then fluorouracil 400 mg/m^2 administered as an IV bolus, then 2400 mg/m^2 administered as a continuous IV infusion over 46 hours.
Drug: FOLFIRI — Following administration of bevacizumab, patients received irinotecan 180 mg/m^2 IV administered over 90 minutes concurrently with folinic acid 400 mg/m^2 (d,I-racemic form, or 200 mg/m^2 I-isomer form) administered IV over 120 minutes, then fluorouracil 400 mg/m^2 administered as an IV bolus, then fluorouracil 2400 mg/m^2 administered as a continuous IV infusion over 46 hours.

SUMMARY:
This was a randomized, placebo-controlled, double-blind study of vismodegib (GDC-0449) added to biochemotherapy standard-of-care regimens for metastatic colorectal cancer (CRC), with treatment until disease progression. Patients received either FOLFOX (FOL=leucovorin calcium [folinic acid], F=fluorouracil, OX=oxaliplatin) or FOLFIRI (FOL=leucovorin calcium [folinic acid] F=fluorouracil, IRI=irinotecan hydrochloride) chemotherapy with bevacizumab. The decision of which regimen (FOLFOX or FOLFIRI) to use was made by the treating physician and patient. Patients were randomized to receive vismodegib or placebo and were stratified based on the chemotherapy regimen chosen and whether or not Response Evaluation Criteria in Solid Tumors (RECIST) measurable disease was present at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed metastatic colorectal cancer (CRC)
* Representative tumor specimens in paraffin blocks (preferred) or at least 15 unstained slides, with an associated pathology report, must be confirmed to be available and requested at any time prior to entry of study
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematopoetic capacity
* Adequate hepatic function
* Adequate renal function
* Use of an effective method of barrier contraception (for women of childbearing potential)
* Signed informed consent

Exclusion Criteria:

* Prior chemotherapy for metastatic CRC or adjuvant chemotherapy for CRC within the prior 6 months
* Clinically suspected or confirmed CNS metastases or carcinomatous meningitis
* Major surgical procedure within 4 weeks prior to the first day of treatment in this study (Day 1)
* Pelvic radiation within 2 weeks prior to Day 1
* Wound dehiscence requiring intervention, gastrointestinal perforation, or bowel obstruction
* Pregnancy or lactation
* Uncontrolled medical illnesses including the following: Infection requiring intravenous (IV) antibiotics, congestive heart failure not controlled with medication, hypertension not controlled with medication
* Thromboembolic disease
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Low, M.D., Ph.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Started | 98 | 101
Completed | 6 | 18
Not Completed | 92 | 83
Not completed — Adverse Event | 4 | 4
Not completed — Death | 6 | 3
Not completed — Physician decision to withdraw patient | 15 | 9
Not completed — Subject decision to withdraw | 15 | 11
Not completed — Disease progression - radiographic | 41 | 51
Not completed — Disease progression - clinical | 8 | 3
Not completed — Reason for discontinuation not available | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib | Total
Number analyzed (Participants) | 98 | 101 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.4) | 60.4 (11.0) | 60.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 46 | 85
  Male | 59 | 55 | 114

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from randomization to the earlier of documented disease progression (PD) or death from any cause. PD: At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since treatment started, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions. For patients without measurable disease, PD was defined as an increase in the size of a lesion to one that is measurable or unequivocal progression of a non-target lesion.
Time Frame: From first treatment through the data cut-off date of March 15, 2010, up to 90 weeks
Population: Intent-to-treat patient population: All randomized patients.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Number analyzed (Participants) | 98 | 101
Months | 9.3 [7.98 to 10.51] | 10.1 [9.43 to 11.33]

2. Secondary Outcome: Progression-free Survival (PFS) in Patients With Various Degrees of Hedgehog Antigen Tumor Expression
Description: Indian + Sonic Hedgehog antigen expression was measured by quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) from archival tumor tissue taken from each patient prior to enrollment in the study. Results are reported in 3 categories; the 33% of patients with the lowest level of expression, the 35% of patients with a middle level of expression, and the 32% of patients with the highest level of expression. PFS was defined as the time between randomization and disease progression, as confirmed by radiography, or death for any reason.
Time Frame: From first treatment through the data cut-off date of March 15, 2010, up to 90 weeks
Population: Intent-to-treat patient population: All randomized patients. Tissue for evaluation was only available for 64 patients in the vismodegib group and 75 patients in the placebo group.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Vismodegib 150 mg | Placebo to Vismodegib
Number analyzed (Participants) | 64 | 75
Months
  ≤ 33%, n=(16,30) | 9.2 [3.6 to 15.9] | 9.4 [7.0 to 11.3]
  33% - 67%, n=(18,28) | 7.4 [5.8 to 8.2] | 11.3 [7.1 to 15.8]
  > 67%, n=(30,17) | 10.7 [7.9 to 11.5] | 14.4 [5.3 to NA] — The upper limit of the confidence interval could not be estimated due to sparse data above the median.

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded starting at the time of informed consent until 45 days after the last dose of treatment or after the initiation of new anti-tumor therapy, whichever was earlier, up to 124 weeks.
Description: Adverse events were reported for the safety-evaluable population, which was defined as all patients who received at least one dose of investigational drug treatment.
Groups:
- Placebo With FOLFOX+Bevacizumab; Placebo With FOLFIRI+Bevacizumab: Placebo will be administered beginning on Cycle 1, Day 3 once daily by oral dosing. For Cycles 2 and beyond, placebo will be administered once daily beginning on Day 1.
- Vismodegib (GDC-0449) With FOLFOX+Bevacizumab; Vismodegib (GDC-0449) With FOLFIRI+Bevacizumab: GDC-0449 (150 mg) will be administered beginning on Cycle 1, Day 3 once daily by oral dosing. For Cycles 2 and beyond, GDC-0449 will be administered once daily beginning on Day 1.
Arm/Group | Placebo With FOLFOX+Bevacizumab | Vismodegib (GDC-0449) With FOLFOX+Bevacizumab | Placebo With FOLFIRI+Bevacizumab | Vismodegib (GDC-0449) With FOLFIRI+Bevacizumab
Serious Adverse Events (participants affected / at risk) | 21/62 | 29/61 | 9/36 | 18/37
Other Adverse Events (participants affected / at risk) | 62/62 | 61/61 | 36/36 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With FOLFOX+Bevacizumab (N=62) | Vismodegib (GDC-0449) With FOLFOX+Bevacizumab (N=61) | Placebo With FOLFIRI+Bevacizumab (N=36) | Vismodegib (GDC-0449) With FOLFIRI+Bevacizumab (N=37)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 3 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1
Chest Pain (General disorders) | 1 | 1 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Sudden Death (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 1
Breast Infection (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0 | 0
Catheter Site Infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal Abscess (Infections and infestations) | 2 | 0 | 0 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 7 | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 1 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 3 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 4 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Malignant Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With FOLFOX+Bevacizumab (N=62) | Vismodegib (GDC-0449) With FOLFOX+Bevacizumab (N=61) | Placebo With FOLFIRI+Bevacizumab (N=36) | Vismodegib (GDC-0449) With FOLFIRI+Bevacizumab (N=37)
Neutropenia (Blood and lymphatic system disorders) | 26 | 19 | 13 | 14
Anaemia (Blood and lymphatic system disorders) | 21 | 14 | 11 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 9 | 5 | 2
Leukopenia (Blood and lymphatic system disorders) | 11 | 6 | 6 | 4
Lymphopenia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 1
Lacrimation Increased (Eye disorders) | 2 | 3 | 1 | 6
Nausea (Gastrointestinal disorders) | 40 | 38 | 21 | 23
Diarrhoea (Gastrointestinal disorders) | 36 | 30 | 29 | 22
Vomiting (Gastrointestinal disorders) | 16 | 23 | 15 | 19
Constipation (Gastrointestinal disorders) | 21 | 20 | 13 | 12
Abdominal Pain (Gastrointestinal disorders) | 13 | 12 | 8 | 6
Stomatitis (Gastrointestinal disorders) | 12 | 8 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 9 | 6 | 5 | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 5 | 3 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 4 | 4 | 3
Oral Pain (Gastrointestinal disorders) | 4 | 2 | 1 | 4
Rectal Haemorrhage (Gastrointestinal disorders) | 4 | 4 | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 8 | 3
Dysphagia (Gastrointestinal disorders) | 5 | 2 | 1 | 1
Flatulence (Gastrointestinal disorders) | 4 | 0 | 1 | 2
Proctalgia (Gastrointestinal disorders) | 3 | 1 | 4 | 1
Fatigue (General disorders) | 42 | 40 | 29 | 27
Mucosal Inflammation (General disorders) | 16 | 15 | 8 | 13
Asthenia (General disorders) | 6 | 10 | 3 | 9
Temperature Intolerance (General disorders) | 20 | 12 | 0 | 1
Pyrexia (General disorders) | 3 | 7 | 6 | 5
Chest Pain (General disorders) | 3 | 5 | 2 | 4
Oedema Peripheral (General disorders) | 3 | 6 | 7 | 2
Pain (General disorders) | 3 | 5 | 3 | 0
Chills (General disorders) | 4 | 3 | 1 | 1
Seasonal Allergy (Immune system disorders) | 2 | 0 | 4 | 0
Urinary Tract Infection (Infections and infestations) | 5 | 11 | 8 | 5
Sinusitis (Infections and infestations) | 1 | 5 | 3 | 4
Oral Candidiasis (Infections and infestations) | 0 | 2 | 0 | 3
Pneumonia (Infections and infestations) | 1 | 3 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 3 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 4 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 3
Weight Decreased (Investigations) | 9 | 20 | 4 | 15
Blood Alkaline Phosphatase Increased (Investigations) | 5 | 3 | 2 | 3
Alanine Aminotransferase Increased (Investigations) | 5 | 1 | 2 | 2
Aspartate Aminotransferase Increased (Investigations) | 6 | 1 | 2 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 31 | 10 | 18
Dehydration (Metabolism and nutrition disorders) | 6 | 13 | 3 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 10 | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 8 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 5 | 2 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 7 | 1 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 7 | 4 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 7 | 7 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 6 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 8 | 29 | 1 | 12
Neuropathy Peripheral (Nervous system disorders) | 34 | 19 | 6 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 14 | 20 | 4 | 1
Dizziness (Nervous system disorders) | 10 | 14 | 2 | 3
Headache (Nervous system disorders) | 16 | 9 | 5 | 5
Syncope (Nervous system disorders) | 3 | 4 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 7 | 9 | 5
Anxiety (Psychiatric disorders) | 3 | 4 | 6 | 7
Depression (Psychiatric disorders) | 3 | 6 | 5 | 4
Proteinuria (Renal and urinary disorders) | 9 | 6 | 6 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 16 | 17 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 9 | 6
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 4 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 11 | 9 | 8
Rash (Skin and subcutaneous tissue disorders) | 8 | 6 | 6 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 4 | 6 | 6 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 2 | 4 | 2
Hypertension (Vascular disorders) | 11 | 6 | 5 | 5
Deep Vein Thrombosis (Vascular disorders) | 0 | 6 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.